CLINICAL TRIAL: NCT03504904
Title: Psychological Treatment Targeting Acceptance and Compassion in Chronic Pain Patients: a Randomized Controlled, Internet Delivered, Treatment Trial.
Brief Title: Psychological Treatment Targeting Acceptance and Compassion in Chronic Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other); Örebro University, Sweden (Other); Karlstad University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 214/248
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Chronic Pain; Self-Criticism
Keywords: Chronic pain; Self-criticism; Internet-based treatment; ACT; CFT; Guided self-help; Acceptance; Compassion
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-delivered ACT and CFT (Experimental): 8 week, guided internet- delivered acceptance and commitment therapy (ACT) and compassion focused therapy (CFT)
  Interventions: Behavioral: Internet-Delivered ACT and CFT
- Wait list control group (No Intervention): Wait list control group, received treatment at later point.

INTERVENTIONS:
Behavioral: Internet-Delivered ACT and CFT — An 8-week internet-based intervention focused on acceptance and compassion. Psychological intervention based on Acceptance and commitment therapy and compassion focused therapy
  Arms: Internet-delivered ACT and CFT

SUMMARY:
This trial is a randomized controlled study aiming to investigate the effect of an 8-week internet-based intervention focused on acceptance and compassion or a wait-list control group. Primary treatments outcomes are Chronic Pain Acceptance Questionnaire (CPAQ), Self-Compassion Scale (SCS) and Pain Disability index (PDI). Secondary outcomes were Montgomery Åsberg Depression Rating Scale (MADRS-S), Anxiety sensitivity index (ASI), Quality of Life Inventory (QOLI), Multidimensional Pain Inventory (MPI) and Perseverative Thinking Questionnaire (PTQ). A six month follow-up was conducted. Findings showed significantly greater levels of acceptance (CPAQ), self-compassion (SCS) and reduction in activity limitation (PDI) measured with the primary outcomes for the treatment group after the intervention with effect sizes raging from small to moderate and these results were maintained at six-month follow-up.

DETAILED DESCRIPTION:
The purpose of this study was to explore if a psychological treatment fusing ACT and CFT principles and therapeutic techniques could improve outcome in chronic pain patients with high levels of self-criticism in comparison to a wait-list control group. The treatment was delivered via the internet, guided by trained professional. Internet delivered cognitive behavior therapy (CBT) and ACT treatments have shown similar efficacy as compared to face-to-face treatments in a variety of problem areas and across a large range of outcomes. Participants were recruited from a clinical setting. The treatment program consisted of eight sections and was based on a manual based on ACT developed for chronic pain (Buhrman et al., 2013) and a CFT-manual for chronic pain.

Following a screening interview participants deemed eligible were asked to complete an assessment battery online. All correspondence concerning treatment was held through a web portal including the online questionnaires and a secure e-mail service. The system handled security issues with two factor authentication. The participants logged in with electronic identification which is a secure service used by banks and in clinical settings.

Measures were obtained pre- and post- intervention and administered via the internet. A sixth month follow-up of the treatment group was administered. Mediation measures were also obtained.

ELIGIBILITY:
Inclusion Criteria:

* have experienced pain for more than three months,
* have been medically investigated (within the past year)
* be at least 18 years of age
* have regular access to a computer and the internet
* reported self-criticism measured with the Self-Compassion Scale.

Exclusion Criteria:

* planned surgery
* ongoing medical investigation that could impede participation in the study,
* suffering from acute physical or psychological conditions,
* very severe symptoms of depression (i.e., defined as a score of >2 on item 9 on MADRS-S and information from telephone screening)
* ongoing psychological treatment,
* not being fluent with the Swedish language since all the material would be in Swedish.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-11-13 (Actual); Primary Completion 2016-01-23 (Actual); Study Completion 2016-01-23 (Actual)

PRIMARY OUTCOMES:
Chronic Pain Acceptance Questionnaire (CPAQ) | At 3, 8 weeks (post-treatment) and 6 months follow-up
  Chronic pain acceptance questionnaire (CPAQ) measures acceptance. The measure consists of two scales; willingness and activity engagement. Items are rated on a scale from 0 (never true) to 6 (always true).Higher scores denote greater activity engagement and pain willingness.The total score is also reported
Self-Compassion Scale (SCS) | At 3, 8 weeks (post-treatment) and 6 months follow-up
  Change from baseline in compassion. The items in Self-Compassion Scale (SCS) are rated on a likert scale from 1(almost never) to 5 (almost always). The scale is divided into six subscales: self-kindness (higher values are considered better), self-judgement (lower values are considered better), common humanity (higher values are considered better), isolation(lower values are considered better), mindfulness (highervalues are considered better) and over-identified (lower values are considered better).Higher scores in the total scale indicate higher levels of compassion. l scale.Results can be presented for the different subclass or a total score. To compute a total self-compassion score, you reverse the negative scales items (self-judgment, isolation, and over-identification ) before computing the grand mean. Subscale scores are computed by calculating the mean of subscale item responses. Higher scores indicate higher levels of self-compassion. A total score can also be reported.
Pain Disability index (PDI) | At 8 weeks (post-treatment) and 6 months follow-up
  Change from baseline in disability. It measures the degree to which pain. Every item score can range from 0 (no interference) to 10 (total interference). The total PDI score can range from 0 to 70, a higher score indicating more interference interferes with functioning across a range of activities.

SECONDARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale (MADRS-S) | At 8 weeks (post-treatment) and 6 months follow-up
  Change from baseline in depression.The respondents rate their symptoms on a scale that ranges from 0 to 6, where a higher value indicates a higher level of depressive symptoms. The score can range from 0-54, higher scores indicate more severe depressive symptoms e.g. a score >35 indicates a severe depression. The questionnaire includes questions on the following symptoms 1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts
Anxiety sensitivity index (ASI) | At 8 weeks (post-treatment) and 6 months follow-up
  Change from baseline in anxiety sensitivity. The ASI total score is the sum of the responses across the 16 items. Higher scores indicate level of anxiety.
Quality of Life Inventory (QOLI) | At 8 weeks (post-treatment) and 6 months follow-up
  Change from baseline in quality of life. The assessment yields an overall score and profile in 16 areas of life; health, self-esteem, goals and values, money, work, play, learning, creativity, helping, love, friends, children, relatives, home, neighbourhood, and community. Higher scores indicate higher level of quality of life.
Multidimensional Pain Inventory (MPI) | At 8 weeks (post-treatment) and 6 months follow-up
  Change from baseline in different pain dimensions. The Swedish version of MPI (MPI-S) consists of 34 items divided into 8 scales. The values on each scale ranges from 0.0-6.0. In some scales higher levels indicate more negative consequences of pain e.g the pain intensity and in other higher scores are positive e.g. life control.
Perseverative Thinking Questionnaire (PTQ) | At 3, 8 weeks (post-treatment) and 6 months follow-up
  Change from baseline in perseverative thinking. It consist of 15 items, every statements are assessed in a likert scale that ranges from 0 (never) to 4 (almost always) and these are divided in three subscales. The subscales are Core characteristics of repetitive negative thinking (RNT), Perceived unproductiveness and Mental capacity. Lower scores indicate lower levels of preservative thinking.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Buhrman, PhD, Principal Investigator — Uppsala University; Katja Boersma, PhD, Study Chair — Örebro University, Sweden; Maria Tillfors, PhD, Study Chair — Karlstad University; Fredrik Holländare, PhD, Study Chair — Örebro University, Sweden
Locations (1):
- Department of Psychology, Uppsala University, Uppsala, Uppland, Sweden

IPD SHARING:
Plan to Share IPD: No